CLINICAL TRIAL: NCT03452527
Title: A Phase 2 Randomized, Open-Label, Multicenter Study Evaluating Administration of Repeated Intravitreal Doses of ICON-1 in Patients With Choroidal Neovascularization Secondary to Age-related Macular Degeneration
Brief Title: Open-Label Study of Intravitreal ICON-1 in Patients With Choroidal Neovascularization Secondary to Age-related Macular Degeneration (AMD)
Acronym: DECO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business Reasons
Sponsor: Iconic Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IT-004
Record Dates: First submitted 2018-02-26; First posted 2018-03-02 (Actual); Results first posted 2021-03-15 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2020-11

CONDITIONS: Choroidal Neovascularization; Wet Macular Degeneration
MeSH Terms: conditions — Choroidal Neovascularization; Wet Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ICON-1 maintenance therapy (Experimental): ICON-1 maintenance therapy after initial aflibercept treatment
  Interventions: Biological: ICON-1; Biological: aflibercept
- ICON-1 combination therapy (Experimental): ICON-1 combination therapy with aflibercept treatment
  Interventions: Biological: ICON-1; Biological: aflibercept

INTERVENTIONS:
Biological: ICON-1 — ICON-1 0.6 mg by intravitreal injection
  Other Names: human Immuno-conjugate 1
Biological: aflibercept — aflibercept 2 mg by intravitreal injection
  Other Names: Eylea®

SUMMARY:
The purpose of this study is to evaluate the safety and effects of repeated intravitreal injections of ICON-1 0.6 mg administered as maintenance therapy or in combination with aflibercept in patients with wet macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Males or females of any race, ≥50 years of age
* Active primary CNV secondary to AMD in the study eye

Exclusion Criteria:

* Any prior treatment of CNV or advanced AMD in the study eye, except for dietary supplements or vitamins
* Any intraocular or ocular surface surgery (including cataract surgery and laser procedures) in the study eye within 3 months
* Vitrectomy in the study eye

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2019-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Burian, MD, Study Director — Iconic Therapeutics, Inc.
Locations (8):
- United States (8):
  - Site 2, Beverly Hills, California
  - Site 8, Santa Ana, California
  - Site 7, Syracuse, New York
  - Site 3, Ashland, Oregon
  - Site 6, Philadelphia, Pennsylvania
  - Site 1, Austin, Texas
  - Site 4, McAllen, Texas
  - Site 5, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ICON-1 Maintenance Therapy | ICON-1 Combination Therapy
Started | 7 | 8
Completed | 4 | 4
Not Completed | 3 | 4
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Study Terminated | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ICON-1 Maintenance Therapy | ICON-1 Combination Therapy | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Customized [Count of Participants; unit: Participants]
  50 to <65 Years | 0 | 1 | 1
  65 to<75 Years | 1 | 2 | 3
  75 to <85 | 3 | 3 | 6
  85 Years or older | 3 | 2 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 2 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 7 | 6 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 8 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Choroidal Neovascularization (CNV) Over Time
Description: Mean change from baseline in CNV area in the study eye
Time Frame: Month 9
Population: The change in choroidal neovascularization by OCT-A, reported as assessed by the investigators. The changes did not correlate with the change in choroidal neovascularization by FA and therefore further analysis was not performed.
Measure: Number; unit: participants
Arm/Group | ICON-1 Maintenance Therapy | ICON-1 Combination Therapy
Number analyzed (Participants) | 5 | 8
participants
  CNV Size-Smaller | 2 | 5
  CNV Size-No Change | 2 | 2
  CNV Size- Larger | 0 | 1
  CNV Size-Cannot Grade | 1 | 0

2. Secondary Outcome: Change in Best Corrected Visual Acuity (BCVA) Over Time
Description: Mean change from baseline in BCVA letter score in the study eye
Time Frame: Month 9
Population: Due to the small sample size and early termination of the study conclusions can not be accurately made from the available data.
Measure: Mean (Full Range); unit: Letters
Arm/Group | ICON-1 Maintenance Therapy | ICON-1 Combination Therapy
Number analyzed (Participants) | 6 | 8
Letters | 1 [-2 to 7] | 0 [-3 to 5]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected during the study period which included the study period plus 30 days after the last dose for a total period of approximately 10 months for patients who completed the trial.
Arm/Group | ICON-1 Maintenance Therapy | ICON-1 Combination Therapy
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 2/7 | 1/8
Other Adverse Events (participants affected / at risk) | 6/7 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ICON-1 Maintenance Therapy (N=7) | ICON-1 Combination Therapy (N=8)
Transient Ischemic Attach (TIA) (Vascular disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Metabolic Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ICON-1 Maintenance Therapy (N=7) | ICON-1 Combination Therapy (N=8)
Macular Fibrosis (Eye disorders) | 1 (1) | 1 (1)
Photopsia (Eye disorders) | 1 (1) | 1 (1)
Retinal Haemorrhage (Eye disorders) | 1 (1) | 1 (1)
Subretinal Fluid (Eye disorders) | 0 (0) | 2 (2)
Choroidal Neovascularization (Eye disorders) | 0 (0) | 1 (1)
Conjunctival Haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Detachment of Retinal Pigment Epithelium (Eye disorders) | 0 (0) | 1 (1)
Dry Age Related Macular Degeneration (Eye disorders) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Eyelids Pruritus (Eye disorders) | 0 (0) | 1 (1)
Lacrimation Increased (Eye disorders) | 1 (1) | 0 (0)
Macular Oedema (Eye disorders) | 0 (0) | 1 (1)
Metamorphopsia (Eye disorders) | 1 (1) | 0 (0)
Optic Ischaemic Neuropathy (Eye disorders) | 0 (0) | 1 (1)
Retinal Depigmentation (Eye disorders) | 0 (0) | 1 (1)
Retinal Pigment Epithelial Tear (Eye disorders) | 1 (1) | 0 (0)
Visual Acuity Reduced (Eye disorders) | 1 (1) | 0 (0)
Visual lmpairement (Eye disorders) | 1 (1) | 0 (0)
Vitreous Detachment (Eye disorders) | 0 (0) | 1 (1)
Vitreous Haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Intraocular Pressure Increased (Eye disorders) | 1 (1) | 2 (2)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Eye disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Drug Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 2 (2)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Genital Herpes (Infections and infestations) | 0 (0) | 1 (1)
Wound Infection (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-19): https://cdn.clinicaltrials.gov/large-docs/27/NCT03452527/Prot_SAP_000.pdf